CLINICAL TRIAL: NCT06383104
Title: Combination of Myofascial Techniques and Proprioceptive Neuromuscular Facilitation in the Clinical and Functional Improvement of Patients With Systemic Lupus Erythematosus. Randomised Clinical Study
Brief Title: Myofascial Techniques and Proprioceptive Neuromuscular Facilitation in Patients With Systemic Lupus Erythematosus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MyoLupus
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-04

CONDITIONS: System; Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Physiotherapy; Joint pain; Range of motion; Functionality; Balance; Fatigue
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthralgia; Fatigue | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention period will last 4 weeks, with a periodicity of 2 weekly sessions of 50 minutes each. The intervention of the experimental group will consist of a protocol using myofascial and proprioceptive neuromuscular facilitation techniques.
  Interventions: Other: Intervention
- Control group (No Intervention): Patients included in the control group will not receive any intervention, maintaining their activities of daily living in the same way as before the study.

INTERVENTIONS:
Other: Intervention — Three myofascial release techniques will be performed with low load and long duration stretching to the myofascial complex to restore optimal length, decrease pain and improve function. In the development of the deep myofascial techniques, respiratory synchronisation with the patient will be performed. Proprioceptive neuromuscular facilitation techniques will be performed by executing diagonal spiral movements against resistance, several times, through a full range of motion. Three sets of three repetitions with 6-second contractions and a 30-second rest between sets shall be performed.
  Arms: Experimental group

SUMMARY:
Introduction. Systemic lupus erythematosus is an autoimmune disease. The musculoskeletal system is affected in 90% of patients. The most common manifestations are myalgias, arthralgias and arthritis.

Objective. To analyse the efficacy of an intervention using myofascial techniques and proprioceptive neuromuscular facilitation in patients with systemic lupus erythematosus.

Methods. Randomised clinical study with 20 patients with systemic lupus erythematosus, randomised to an experimental and control group. The intervention will last 4 weeks, with a periodicity of 2 weekly sessions of 50 minutes each. The intervention of the experimental group will consist of a protocol using myofascial and proprioceptive neuromuscular facilitation techniques.

Expected results. Improvement of knee and ankle pain intensity, functional capacity, basic mobility skills, strength, balance, agility and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age
* With a medical diagnosis of systemic lupus erythematosus
* Who sign the informed consent form.

Exclusion Criteria:

* Patients with fever or acute phlebitis.
* Patients with recent lower limb fractures
* Amputees and people with neurological or cognitive impairments that prevent them from correctly understanding the questionnaires and performing the guided techniques.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline joint pain after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  The intensity of knee and ankle pain shall be measured with the visual analogue scale. This instrument has an excellent test-retest reliability. This measurement scale consists of an unnumbered 10 cm line, where the patient is asked to indicate the perception of pain in the knee and ankle joints in the last week. The scale ranges from 0 to 10, where 0 indicates no pain at all and 10 indicates maximum perceived pain.

SECONDARY OUTCOMES:
Change from baseline functional capacity after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Functionality of the lower limbs will be measured with the 2-Minute Walking Test. Functional capacity to exercise will be assessed by this modified version of the 6-minute version. This instrument has shown excellent test-retest reliability. This test will be performed in a closed corridor, with a length of 30 m delimited between cones. Subsequently, they shall be instructed to walk around the circuit around the cones as fast as possible, but without running, for 2 minutes. The distance covered at the end of the 2 minutes, in metres, shall be recorded by the assessor.
Change from baseline functionality after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  The Timed Up and Go Functionality Test will assess basic mobility skills, strength, balance and agility. This instrument can help predict an individual's risk of falls and other adverse outcomes. This test has shown excellent intra-rater reliability. This test measures the time it takes a patient to get up from an armchair (without using the arms to get up), walk to a line on the floor 3 m away, turn around, and return to the chair and sit down. The unit of measurement is seconds
Change from baseline joint pain after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Fatigue will be assessed using the Fatigue Assessment Scale. This scale provides information on physical and psychological aspects of fatigue. The reliability of this scale is high. This instrument is a self-report questionnaire consisting of 10 items with a 5-point Likert response scale ranging from "1=never to "5=Always". Five items reflect the physical component and five reflect the psychological component. The score range of the scale is 10-50, where the higher the score, the greater the degree of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No